CLINICAL TRIAL: NCT02763020
Title: Postprandial Glycemic Response to Polyphenol-fortified Snack Bars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15-28-HC
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Blood Sugar Response
Keywords: high glycemic index, polyphenols, blood glucose, satiety
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Food bar without fruit (Placebo Comparator): snack bar without fruit
  Interventions: Other: placebo
- Food bar with cranberry extract (0.5%) (Experimental): Snack bar with cranberry extract (0.5% total weight)
  Interventions: Other: Fruit extracts high in polyphenols
- Food bar with cranberry extract (1.0%) (Experimental): Snack bar with cranberry extract (1.0% total weight)
  Interventions: Other: Fruit extracts high in polyphenols
- Food bar w/ dried black raspberry (10%) (Experimental): Snack bar with freeze-dried black raspberry(10% total weight)
  Interventions: Other: Fruit extracts high in polyphenols
- Food bar w/ dried black raspberry (20%) (Experimental): Snack bar with freeze-dried black raspberry (20% total weight)
  Interventions: Other: Fruit extracts high in polyphenols

INTERVENTIONS:
Other: Fruit extracts high in polyphenols
  Arms: Food bar w/ dried black raspberry (10%); Food bar w/ dried black raspberry (20%); Food bar with cranberry extract (0.5%); Food bar with cranberry extract (1.0%)
Other: placebo
  Arms: Food bar without fruit

SUMMARY:
Consuming plant chemicals (e.g., polyphenols) may have beneficial effects on human health that, if confirmed, may warrant inclusion in combat rations. Ration developers would like to determine whether the fortification of a high sugar food item with a polyphenol-rich freeze-dried fruit and/or a fruit extract improves blood sugar response and promotes other positive physiological changes (e.g., satiety) in a dose-response manner. This study will test four different types of snack bar with various polyphenol doses, and compare blood response to a snack bar without polyphenols.

DETAILED DESCRIPTION:
High glycemic index (GI) foods generally contain simple sugars and/or highly processed and refined carbohydrates (e.g., instant oatmeal and white bread). These foods are rapidly digested, which raises blood glucose and insulin to higher concentrations and more rapidly compared to low GI food items. In some situations, it is advantageous to consume high glycemic response food items to promote recovery from intense exercise/work. However, there is some suggestion that low/moderate-GI foods may better maintain glucose levels and enhance performance if consumed before and during prolonged exercise. Further, impaired blood glucose regulation (e.g., that can occur with chronic intake of high GI foods) may stimulate the development of oxidative stress, inflammation, dyslipidemia, insulin resistance, and diabetes; and, it is associated with changes in body weight due to stimulating hunger and excessive food intake. These negative consequences are concerning, given the prevalence of overweight/obesity and comorbidities (including metabolic syndrome) within the Department of Defense (DoD). Polyphenols are a heterogeneous group of phytochemicals that are found in plant-based foods; and they have antioxidant and anti-inflammatory properties that may ultimately help protect against chronic diseases, such as cancer and cardiometabolic disease. Berry polyphenols are predominantly comprised of proanthocyanidins and/or ellagitannins (collectively referred to as "tannins"); and, berries have been shown to promote glycemic control when consumed with a high-carbohydrate containing food item. These beneficial health effects may warrant polyphenol fortification of combat rations and Garrison food items. For example, Natick Soldier Research, Development and Engineering Center's (NSRDEC) Combat Feeding Directorate demonstrated that tannins extracted from berries effectively inhibits the activity of enzymes that metabolize starch in vitro, an underlying mechanism for slowing starch digestion in vivo. However, whether consumption of a high GI food item containing polyphenol-rich freeze-dried fruit and/or fruit extracts improves glucose control, reduces oxidative stress, and promotes satiety in human volunteers is unknown. In this randomized, cross-over, placebo-controlled, dose-response trial, at least 20 civilian and/or military personnel will be asked to consume one of five food items during separate trials: 1) a high glycemic snack bar (control) without any fruit ingredients; 2) a high glycemic snack bar with cranberry extract (0.5% total weight); 3) a high glycemic snack bar with cranberry extract (1% total weight); 4) a high glycemic bar with freeze-dried black raspberries (10% total weight); and, 5) a high glycemic snack bar with freeze-dried black raspberries (20% total weight). Serial blood sampling to measure acute changes in circulating glucose, insulin, gastrointestinal hormones and biomarkers of oxidative stress and satiety will occur at baseline and for three hours after consumption of each food. Appetite will also be assessed at an ad libitum meal after the three hour period. The only known risks, which this study presents to participants, are those associated with venous catheter placement. The fruit concentrates for the present study are either commercially available (black raspberry powders) or used as an ingredient to boost the phenolic content of commercial items (cranberry extract). The results will help determine whether fortifying high glycemic food items with polyphenols may benefit the Warfighter in the ration- or Garrison-feeding environment.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers who are stationed with USARIEM, NSRDEC or the U.S. Army Natick Soldier Center pool of military participants, or any civilians will be invited to participate in this study.

Exclusion Criteria:

* Potential participants will be excluded from participation if they: are under the age of 18 or over the age of 39 (i.e. insulin sensitivity declines with age, hence the upper age limit of 39 years); have a pre-existing liver disease, history of alcoholism or typically consume more than 4 alcoholic beverages daily or 6 on one occasion more than once a month within the past 6 months; have impaired glucose metabolism due to diabetes, pre-diabetes, galactosemia, hereditary fructose intolerance or glycogen storage disease; have thyroid disease; have a bleeding disorder (e.g., von Willebrand Disease, hemophilia) or are being treated with medication that will impair blood clotting; have a history of GI-related conditions that may impact glucose absorption (e.g., Crohn's disease, ulcerative colitis, Celiac's disease or gluten sensitivity, bariatric surgery or gastroparesis); are taking any medications affecting carbohydrate metabolism (e.g., insulin or oral diabetes medications); and/or, have an allergy or aversion to any of the test foods.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
blood glucose concentrations | fasting and post-prandial (every 15 minutes for the first hour and every half hour for the last two hours)

SECONDARY OUTCOMES:
gut hormones | fasting and post-prandial (every 15 minutes for the first hour and every half hour for the last two hours)
blood concentration of phenolic acids | fasting, post-prandial 60 minutes, 120 minutes and 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Smith, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No